CLINICAL TRIAL: NCT05073211
Title: A Randomized Split-face Study of Photodynamic Therapy With St. John's Wort Versus Indole-3-acetic Acid for the Treatment of Acne
Brief Title: St. John's Wort Photodynamic Therapy
Acronym: SJWPDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Shin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1906547-003
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: a double-blind split-face randomized controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SJW-PDT (Experimental): Participants were randomized to receive either the SJW extract or IAA on each split-face. The SJW extract (DR-Light complexTM; Genicos Co., Ltd, Cheongju, Korea) consisted of 70% 1, 3-butylene glycol, and 0.1% hypericin as active ingredients. After cleansing the face gently, participants applied 1.5 ml of 0.5% SJW extract on one half of the face and 1.5 ml of 0.015% IAA (AC gel®; Wellskin, Seoul, Korea) on the other half of the face for 10 minutes under occlusion.
  Interventions: Procedure: PDT
- IAA-PDT (Active Comparator): Participants were randomized to receive either the SJW extract or IAA on each split-face. The SJW extract (DR-Light complexTM; Genicos Co., Ltd, Cheongju, Korea) consisted of 70% 1, 3-butylene glycol, and 0.1% hypericin as active ingredients. After cleansing the face gently, participants applied 1.5 ml of 0.5% SJW extract on one half of the face and 1.5 ml of 0.015% IAA (AC gel®; Wellskin, Seoul, Korea) on the other half of the face for 10 minutes under occlusion.
  Interventions: Procedure: PDT

INTERVENTIONS:
Procedure: PDT — A 630 nm red light and a 520 nm green light of the light-emitting diode (LED) device (Nouvo-GB®) with an intensity of 35 mW⁄cm2 was simultaneously illuminated for 10 minutes (a total light dose of 21 J/cm2). Participants received a total of four treatments at 1-week intervals and were followed up 1 and 4 weeks after the last treatment.

SUMMARY:
The investigators aimed to evaluated the efficacy and safety of SJW-PDT compared to indole-3-acetic acid (IAA)-PDT in the treatment of acne. The investigators also investigated the skin rejuvenating effects of SJW-PDT.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate facial acne
* between 25 and 60 years old

Exclusion Criteria:

* history of oral retinoid treatment with the past 6 months
* history of oral antibiotics, topical acne treatment, or skin rejuvenation treatment such as lasers and chemical peeling within the month before the start of the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
acne lesions | 1 and 4 weeks after the last treatment
  change in the number of acne lesions after the treatment

SECONDARY OUTCOMES:
sebum secretion rate (μg/cm2) | 1 and 4 weeks after the last treatment
  Sebum secretion rate was measured with Sebumeter SM 815®.

OTHER OUTCOMES:
erythema index (arbitrary unit) | 1 and 4 weeks after the last treatment
  The erythema index (EI) was measured with Mexameter MX 1® (Courage & Khazaka)
skin texture, wrinkles (arbitrary unit) | 1 and 4 weeks after the last treatment
  The skin texture and wrinkles were measured with an Antera 3D® camera (Miravex Limited, Dublin, Ireland).

CONTACTS AND LOCATIONS:
Overall Officials: Jung Won Shin, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BR, Kim M, Na JI, Huh CH, Shin JW. A Randomized Split-Face Study of Photodynamic Therapy With St. John's Wort and Indole-3-Acetic Acid for the Treatment of Acne. Dermatol Surg. 2023 May 1;49(5):483-488. doi: 10.1097/DSS.0000000000003742. Epub 2023 Mar 21. PMID 36946749